CLINICAL TRIAL: NCT02731664
Title: GLP-1 Inhibits Prandial Antro-duodeno-jejunal Motility in Humans: Native GLP-1 Compared With Analogue ROSE-010 in Vitro
Brief Title: GLP-1 Inhibits Prandial Antro-duodeno-jejunal Motility in Humans
Acronym: GLPMOT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Hellström, Professor, Uppsala University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PRANDMOTGLP
Record Dates: First submitted 2016-03-06; First posted 2016-04-07 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Irritable bowel syndrome; Functional dyspepsia; Gastric emptying; Gastrointestinal peptide hormones
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLP-1 (Experimental): Intravenous infusion of GLP-1 at 0.7 and 1.2 mol/kg per minute
  Interventions: Biological: GLP-1
- Control (Placebo Comparator): Intravenous saline
  Interventions: Biological: Intravenous saline

INTERVENTIONS:
Biological: GLP-1 — Intravenous infusion of GLP-1
  Other Names: Glucagon-like peptide-1
  Arms: GLP-1
Biological: Intravenous saline — Control
  Arms: Control

SUMMARY:
The inhibitory effect of low dose GLP-1 is investigated on prandial motility of the stomach, duodenum and jejunum in vivo in humans. Supplementary in vitro studies on the mechanism of action of the GLP-1 inhibition of motility as carried out on muscle strips from the upper gastrointestinal tract in man.

DETAILED DESCRIPTION:
Twelve healthy volunteers will undergo antroduodenojejunal manometry. Baseline recording with infusion of saline for 1 hour is compared with infusion of GLP-1 0.7 and 1.2 pmol per kg minute for another 1 hour. Plasma GLP-1 and GLP-2 is measured by RIA. Responses to GLP-1 will be measured after food intake as prandial response to GLP-1. The outcome will be evaluated as change in motility index from baseline to meal-stimulated conditions and during influence of GLP-1. Further in vitro studies of gastrointestinal muscle strips, precontracted with bethanechol or electric field stimulation, are planned to investigate the response to GLP-1 or GLP-1 analogue ROSE-010. GLP-1 and GLP-2 receptor immunoreactivity is localized by immunohistochemistry. Receptor mediated mechanisms are studied with GLP-1 receptor blocker exendin(9-39)amide, nitro-monomethyl arginine to block nitric oxide synthase and tetrodotoxin to block sodium channels and nerve conduction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers over 18 years of age.

Exclusion Criteria:

* Any medical condition.
* Any drug treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Motility index (measure of contraction amplitude x duration; area for mmHg x sec) | 60 minutes
  Inhibition of prandially increased motility index (motor activity in the antrum and upper small intestine).

SECONDARY OUTCOMES:
Smooth muscle relaxation induced by GLP-1 | 6 hours
  Separate experiments in vitro: GLP-1-induced inhibition of bethanechol-stimulated smooth muscle strips to characterize GLP-1's pharmacological action.
Presence of GLP-1 and GLP-2 receptors in gastric and small bowel tissue | 1 day
  Separate experiments in vitro: Antibody staining of gastric and small bowel tissue for receptors of GLP-1 and GLP-2

CONTACTS AND LOCATIONS:
Overall Officials: Per M. Hellström, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
On request.

REFERENCES:
- [Background] Edholm T, Degerblad M, Gryback P, Hilsted L, Holst JJ, Jacobsson H, Efendic S, Schmidt PT, Hellstrom PM. Differential incretin effects of GIP and GLP-1 on gastric emptying, appetite, and insulin-glucose homeostasis. Neurogastroenterol Motil. 2010 Nov;22(11):1191-200, e315. doi: 10.1111/j.1365-2982.2010.01554.x. PMID 20584260
- [Background] Hellstrom PM, Hein J, Bytzer P, Bjornsson E, Kristensen J, Schambye H. Clinical trial: the glucagon-like peptide-1 analogue ROSE-010 for management of acute pain in patients with irritable bowel syndrome: a randomized, placebo-controlled, double-blind study. Aliment Pharmacol Ther. 2009 Jan;29(2):198-206. doi: 10.1111/j.1365-2036.2008.03870.x. Epub 2008 Oct 10. PMID 18945254
- [Result] Hellstrom PM, Naslund E, Edholm T, Schmidt PT, Kristensen J, Theodorsson E, Holst JJ, Efendic S. GLP-1 suppresses gastrointestinal motility and inhibits the migrating motor complex in healthy subjects and patients with irritable bowel syndrome. Neurogastroenterol Motil. 2008 Jun;20(6):649-59. doi: 10.1111/j.1365-2982.2007.01079.x. Epub 2008 Feb 19. PMID 18298441
- [Derived] Halim MA, Degerblad M, Sundbom M, Karlbom U, Holst JJ, Webb DL, Hellstrom PM. Glucagon-Like Peptide-1 Inhibits Prandial Gastrointestinal Motility Through Myenteric Neuronal Mechanisms in Humans. J Clin Endocrinol Metab. 2018 Feb 1;103(2):575-585. doi: 10.1210/jc.2017-02006. PMID 29177486